CLINICAL TRIAL: NCT00515086
Title: A Phase II Trial of RAD001 in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Study of Everolimus (RAD001) in Patients With Recurrent Glioblastoma Multiforme (GBM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to slow enrollment and protocol-defined stopping rule.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2410
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Results first posted 2011-07-27 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme, GBM, RAD001, RAD
MeSH Terms: conditions — Glioblastoma; Dyschromatosis symmetrica hereditaria 1 | interventions — Everolimus; Surgical Procedures, Operative

ARMS (4):
- No Surgery (Everolimus 10 mg) (Experimental): Participants with recurrent Glioblastoma Multiforme (GBM) not scheduled to undergo salvage surgical resection, received a daily oral dose of 10 mg Everolimus (RAD001) until evidence of disease progression or toxicity.
  Interventions: Drug: Everolimus
- Everolimus 10 mg + Surgery (Experimental): Participants scheduled to undergo salvage surgical resection received a daily oral dose of 10 mg Everolimus for 7 days prior to surgery, then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
  Interventions: Drug: Everolimus; Procedure: Surgery
- Everolimus 5 mg + Surgery (Experimental): Participants scheduled to undergo salvage surgical resection received a daily oral dose of 5 mg Everolimus for 7 days prior to surgery, then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
  Interventions: Drug: Everolimus; Procedure: Surgery
- Everolimus 0 mg + Surgery (Active Comparator): Participants scheduled to undergo salvage surgical resection received no treatment with Everolimus prior to surgery, then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
  Interventions: Drug: Everolimus; Procedure: Surgery

INTERVENTIONS:
Drug: Everolimus — Tablets taken once a day with a full glass of water.
  Other Names: RAD001
Procedure: Surgery — Salvage surgical resection
  Arms: Everolimus 0 mg + Surgery; Everolimus 10 mg + Surgery; Everolimus 5 mg + Surgery

SUMMARY:
This study will define the safety and efficacy of Everolimus (RAD001) administered daily in patients with glioblastoma multiforme (GBM)

DETAILED DESCRIPTION:
This was a multicenter, open label, randomized study of RAD001 dosed daily in patients with recurrent GBM. The study was conducted with 2 parallel groups of patients. Group 1 was designed to study the biological effects of RAD001 in patients scheduled to undergo salvage surgical resection, and Group 2 was to enroll patients who were not scheduled for surgery. Patients in Group 1 were randomly assigned to one of three pre-surgery treatment groups (0, 5 or 10 mg/day RAD001 for 7 days). All patients in Group 2 were to receive a fixed daily dose of 10 mg/day oral RAD001.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Histologically confirmed Glioblastoma Multiforme (GBM)
* Radiographic evidence of disease progression
* Patients must have evaluable contrast enhancing tumor
* Availability of paraffin blocks or unstained pathology slides for biomarker studies
* Karnofsky Performance Status of greater than or equal to 60%

Exclusion Criteria:

* Prior treatment with Mammalian target of rapamycin (mTOR) inhibitor
* History of another malignancy within 3 years
* Cardiac pacemaker
* Ferromagnetic metal implants other than those approves as safe for use in Magnetic resonance imaging (MRI) scanners
* Claustrophobia
* Obesity
* Unstable systemic diseases
* Elevated cholesterol or triglycerides
* Radiation therapy or cytotoxic chemotherapy <=4 weeks prior to study enrollment. Patient must have recovered from the toxic effects of a prior chemotherapy.
* Patients must be off all enzyme inducing anticonvulsants for at least 2 week before study enrollment can occur
* Need for increasing dose of steroids. Patients on a stable or tapering dose of steroids >=7 days were permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke University - Preston Robert Tisch Brain Tumor Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were separated into 2 Groups: Group 1 (Surgery Group) patients were scheduled for salvage surgery and randomly assigned to one of 3 pre-surgery treatment groups: 0, 5 or 10 mg/day Everolimus for 7 days. Group 2 (No Surgery Group) patients were not scheduled for salvage surgery and received 10 mg/day Everolimus.
Groups:
- Everolimus 10 mg + Surgery: Participants scheduled to undergo salvage surgical resection, received a daily oral dose of 10 mg Everolimus for 7 days prior to surgery, then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
- Everolimus 5 mg + Surgery: Participants scheduled to undergo salvage surgical resection, received a daily oral dose of 5 mg Everolimus for 7 days prior to surgery, then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
- Everolimus 0 mg + Surgery: Participants scheduled to undergo salvage surgical resection, received no treatment with Everolimus prior to surgery, then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
Period: Overall Study
Arm/Group | No Surgery (Everolimus 10 mg) | Everolimus 10 mg + Surgery | Everolimus 5 mg + Surgery | Everolimus 0 mg + Surgery
Started | 24 | 6 | 5 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 24 | 6 | 5 | 6
Not completed — Adverse Event | 1 | 1 | 2 | 3
Not completed — Administrative | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 18 | 3 | 3 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Study drug no longer required | 0 | 1 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Surgery (Everolimus 10 mg) | Everolimus 10 mg + Surgery | Everolimus 5 mg + Surgery | Everolimus 0 mg + Surgery | Total
Number analyzed (Participants) | 24 | 6 | 5 | 6 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 5 | 5 | 5 | 29
  >=65 years | 10 | 1 | 0 | 1 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 0 | 4 | 13
  Male | 19 | 2 | 5 | 2 | 28

OUTCOME MEASURES:

1. Primary Outcome: Surgery Group: Percentage Change From the Baseline in S6 Kinase Levels
Description: In the Surgery Group, the primary efficacy assessment was inhibition of Mammalian target of rapamycin (mTOR) as defined as ≥75% S6 phosphorylation. The occurrence of S6 phosphorylation was determined by phosphor-S6 immunohistochemical staining. Tumor cells from the initial surgical resection and from the salvage resection were used for assessments.
Time Frame: Baseline and Day 7-9 (during salvage surgery)
Population: Study was terminated due to slow enrollment.
Measure: Number; unit: Percentage change in S6 kinase
Groups:
- Everolimus 5 mg + Surgery: Participants scheduled to undergo salvage surgical resection, received a daily oral dose of 5 mg Everolimus for 7 days prior to surgery then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
- Everolimus 0 mg + Surgery: Participants scheduled to undergo salvage surgical resection, received no treatment with Everolimus prior to surgery then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
Arm/Group | Everolimus 10 mg + Surgery | Everolimus 5 mg + Surgery | Everolimus 0 mg + Surgery
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: No Surgery Group: Best Overall Tumor Response
Description: The best overall tumor response is reported for participants with 1 previous relapse and participants with ≥2 previous relapses according to the following categories: Complete Response, Partial Response, Stable Disease and Progressive Disease. Gadolinium chelate-enhanced Magnetic Resonance Imaging (MRI) was used for tumor analysis. The objective assessment of tumor response was evaluated at each site by the designated pathologist based on the Neuro-Oncology criteria for Tumor Response for Central Nervous System (CNS) tumors.
Time Frame: First day of treatment to study discontinuation (up to 60 weeks)
Population: No Surgery Group participants from the Intent-to-treat (ITT) population who received at least one dose of study medication.
Measure: Number; unit: Participants
Groups:
- No Surgery (1 Previous Relapse): Participants with recurrent Glioblastoma Multiforme (GBM) with 1 previous relapse not scheduled to undergo salvage surgical resection, received a daily oral dose of 10 mg Everolimus (RAD001) until evidence of disease progression or toxicity.
- No Surgery ( ≥ 2 Previous Relapses): Participants with recurrent Glioblastoma Multiforme with ≥ 2 previous relapses not scheduled to undergo salvage surgical resection, received a daily oral dose of 10 mg Everolimus until evidence of disease progression or toxicity.
Arm/Group | No Surgery (1 Previous Relapse) | No Surgery ( ≥ 2 Previous Relapses)
Number analyzed (Participants) | 12 | 12
Participants
  Complete response + Partial response | 0 | 0
  Complete response | 0 | 0
  Partial response | 0 | 0
  Stable disease | 3 | 6
  Progressive disease | 7 | 6

3. Secondary Outcome: Surgery Group: Blood and Brain Tissue Levels of Everolimus (RAD001)
Time Frame: Baseline and Day 7-9 (Blood samples were collected one day prior to surgery and tissue samples were collected during surgery.)
Population: Study was terminated due to slow enrollment.
Measure: Mean (Standard Deviation); unit: Levels
Arm/Group | Everolimus 10 mg + Surgery | Everolimus 5 mg + Surgery | Everolimus 0 mg + Surgery
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Surgery Group: Progression-free Survival
Description: Progression-free survival (PFS) was assessed using Gadolinium chelate-enhanced Magnetic Resonance Imaging (MRI) and based on the Neuro-Oncology Criteria for Tumor Response for CNS tumors. PFS was measured from the first day of treatment after surgery to disease progression or death and is derived using the Kaplan-Meier method.
Time Frame: After surgery (within 96 hours), Weeks 4 and 8 and then every 8 weeks after restarting treatment until study discontinuation (Up to 28 weeks)
Population: Results for the Surgery Group only include patients with residual tumor following salvage surgery.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Total: All the participants scheduled to undergo salvage surgical resection from three pre-surgery treatment groups (i.e 0, 5 or 10 mg/day (once daily) everolimus X 7 days).
Arm/Group | Everolimus 10 mg + Surgery | Everolimus 5 mg + Surgery | Everolimus 0 mg + Surgery | Total
Number analyzed (Participants) | 6 | 4 | 6 | 16
Weeks | 25.9 [8.7 to 27.1] | 9.1 [5.6 to 14.9] | NA [14.3 to NA] — Because most participants (5) were censored in the no treatment group, the median and upper level limit of the 95% Confidence Interval for Progression-free survival could not be calculated. | 14.9 [9.1 to 27.1]

5. Secondary Outcome: Surgery Group: Biomarkers Phosphatase and Tensin Homolog (PTEN) and Epidermal Growth Factor Receptor (EGFR)
Description: The secondary efficacy assessment was to evaluate the role of PTEN and EGFR pathway status on phosphor-S6. Tumor cells from the initial surgical resection and from the salvage resection were used for assessments. Immunohistochemistry and Fluorescence in-situ hybridization (FISH) were used to assess PTEN and EGFR pathway status.
  Study was terminated due to slow enrollment. Analysis was not possible due to insufficient sample size.
Time Frame: After surgery, week 4, week 8 and every 8 weeks thereafter
Population: Study was terminated due to slow enrollment.
Measure: Mean (Standard Deviation); unit: Levels
Groups:
- Everolimus 10 mg + Surgery: Participants scheduled to undergo salvage surgical resection, received a daily oral dose of 10 mg Everolimus (RAD001) for 7 days prior to surgery then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
- Everolimus 5mg + Surgery: Participants scheduled to undergo salvage surgical resection, received a daily oral dose of 5 mg Everolimus for 7 days prior to surgery then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
Arm/Group | Everolimus 10 mg + Surgery | Everolimus 5mg + Surgery | Everolimus 0 mg + Surgery
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: No Surgery Group: Progression Free Survival
Description: Progression-free survival (PFS) was assessed using Gadolinium chelate-enhanced Magnetic Resonance Imaging (MRI) and based on the Neuro-Oncology Criteria for Tumor Response for CNS tumors. PFS is reported for participants with 1 previous relapse and participants with ≥2 previous relapses. PFS was measured from the first day of treatment to disease progression or death and is derived using the Kaplan-Meier method.
Time Frame: First day of treatment to study discontinuation (up to 60 weeks)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- No Surgery ( ≥ 2 Previous Relapses): Participants with recurrent Glioblastoma Multiforme (GBM) with ≥ 2 previous relapses not scheduled to undergo salvage surgical resection, received a daily oral dose of 10 mg Everolimus until evidence of disease progression or toxicity.
- Total : No Surgery: Total participants enrolled with recurrent glioblastoma multiforme (GBM) who were not scheduled to undergo a planned salvage surgical resection. All participants in this arm were to receive a fixed daily dose of 10 mg/day oral everolimus.
Arm/Group | No Surgery (1 Previous Relapse) | No Surgery ( ≥ 2 Previous Relapses) | Total : No Surgery
Number analyzed (Participants) | 12 | 12 | 24
Weeks | 4.14 [3.7 to 7.0] | 4.14 [3.9 to 12.0] | 4.14 [4.0 to 5.9]

7. Secondary Outcome: Surgery Group: Number of Participants With Adverse Events
Description: The number of participants with any adverse event by System Organ Class. Additional information about Adverse Events can be found in the Adverse Event Section.
Time Frame: First day of treatment to study discontinuation (Up to 28 weeks)
Population: Surgery Group participants from the Safety population who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Everolimus 10 mg + Surgery | Everolimus 5 mg + Surgery | Everolimus 0 mg + Surgery
Number analyzed (Participants) | 6 | 5 | 6
Participants
  Gastrointestinal disorders | 5 | 5 | 3
  Nervous system disorders | 4 | 5 | 5
  General disorders & administration site conditions | 4 | 4 | 5
  Metabolism and nutrition disorders | 6 | 4 | 3
  Blood and lymphatic system disorders | 4 | 2 | 5
  Infections and infestations | 4 | 2 | 3
  Psychiatric disorders | 5 | 3 | 2
  Skin and subcutaneous tissue disorders | 4 | 2 | 2
  Investigations | 3 | 1 | 1
  Injury, poisoning, and procedural complications | 5 | 3 | 0
  Musculoskeletal and connective tissue disorders | 1 | 1 | 2
  Respiratory, thoracic and mediastinal disorders | 0 | 2 | 2
  Renal and urinary disorders | 0 | 1 | 2
  Vascular disorders | 2 | 1 | 2
  Immune system disorders | 1 | 1 | 1
  Eye disorders | 1 | 1 | 0
  Ear and labyrinth disorders | 2 | 0 | 0
  Reproductive system and breast disorders | 0 | 1 | 0
  Cardiac disorders | 0 | 0 | 1
  Endocrine disorders | 1 | 0 | 0
  Surgical and medical procedures | 1 | 0 | 0
  Neoplasms benign, malignant and unspecified | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Everolimus 10 mg + Surgery: Participants scheduled to undergo salvage surgical resection, received a daily oral dose of 10 mg Everolimus for 7 days prior to surgery then after recovery from surgery received a 10 mg daily oral dose of Everolimus until evidence of disease progression or toxicity.
Arm/Group | Everolimus 10 mg + Surgery | Everolimus 5 mg + Surgery | Everolimus 0 mg + Surgery | No Surgery (Everolimus 10 mg)
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/5 | 2/6 | 6/24
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 6/6 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 10 mg + Surgery (N=6) | Everolimus 5 mg + Surgery (N=5) | Everolimus 0 mg + Surgery (N=6) | No Surgery (Everolimus 10 mg) (N=24)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Gait Disturbance (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Bacterial Diarrhoea (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0
Perirectal Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection Staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Pneumocephalus (Nervous system disorders) | 0 | 0 | 0 | 1
intracranial Hypotension (Nervous system disorders) | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 10 mg + Surgery (N=6) | Everolimus 5 mg + Surgery (N=5) | Everolimus 0 mg + Surgery (N=6) | No Surgery (Everolimus 10 mg) (N=24)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 3 | 6
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ear Discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 1 | 0 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 4 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Facial Pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 2 | 8
Irritability (General disorders) | 0 | 0 | 0 | 2
Localised Oedema (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 1 | 3 | 1
Oedema Peripheral (General disorders) | 2 | 0 | 1 | 2
Pain (General disorders) | 0 | 2 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 1 | 1 | 1
Fungal Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0 | 0
Herpes Zoster Oticus (Infections and infestations) | 1 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory Tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0
Upper Respiratory Tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary Tract infection (Infections and infestations) | 1 | 0 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Endotracheal intubation Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Procedural Pain (Injury, poisoning and procedural complications) | 4 | 2 | 0 | 0
Radiation Necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
incision Site Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine Aminotransferase increased (Investigations) | 2 | 1 | 1 | 2
Aspartate Aminotransferase increased (Investigations) | 2 | 0 | 0 | 2
Blood Albumin Decreased (Investigations) | 0 | 0 | 0 | 2
Blood Alkaline Phosphatase increased (Investigations) | 1 | 0 | 1 | 0
Blood Bicarbonate Decreased (Investigations) | 1 | 0 | 0 | 0
Blood Cholesterol increased (Investigations) | 1 | 0 | 0 | 4
Blood Triglycerides increased (Investigations) | 1 | 0 | 0 | 4
Gamma-Glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 0 | 1
Heart Rate increased (Investigations) | 1 | 0 | 0 | 0
Low Density Lipoprotein increased (Investigations) | 0 | 0 | 0 | 3
Oxygen Saturation Decreased (Investigations) | 1 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 1 | 0 | 0 | 3
Protein Total increased (Investigations) | 2 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 3
Weight increased (Investigations) | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 2 | 2 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 3 | 0 | 0 | 0
Brain Oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 2 | 1 | 0 | 1
Depressed Level of Consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 1
Facial Palsy (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 4
Hemianopia (Nervous system disorders) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 1
Hypogeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Memory Impairment (Nervous system disorders) | 1 | 0 | 0 | 1
Mental Impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 3 | 1 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sinus Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Speech Disorder (Nervous system disorders) | 2 | 0 | 1 | 2
Visual Field Defect (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 2
Confusional State (Psychiatric disorders) | 1 | 1 | 1 | 1
Depression (Psychiatric disorders) | 2 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 1
insomnia (Psychiatric disorders) | 2 | 1 | 1 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2
incontinence (Renal and urinary disorders) | 0 | 0 | 2 | 1
Sexual Dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Allergic Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
increased Tendency To Bruise (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Tooth Extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the early termination of this study, the analysis of some of the planned objectives is not included in this clinical study report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or the publication of the trial results in their entirety.